CLINICAL TRIAL: NCT02813590
Title: Ascitic Fluid Microbiome in Liver Cirrhosis
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Medical University of Graz (Other)
Collaborators: CBmed - Center for biomarker research in medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 25-326 ex 12/13
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ascitic Fluid, Microbiota; Microbiota; Sequence Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with liver cirrhosis and with SBP
  Interventions: Other: Ascitic fluid puncture; Other: Skin swaps from puncture side; Other: Stool samples
- Patients with liver cirrhosis and without SBP
  Interventions: Other: Ascitic fluid puncture; Other: Skin swaps from puncture side; Other: Stool samples

INTERVENTIONS:
Other: Ascitic fluid puncture
Other: Skin swaps from puncture side
Other: Stool samples

SUMMARY:
Ascitic fluid microbiome is going to be investigated in this study by using internal transcripted spacer (ITS) and 16S ribosomal RNA (rRNA) polymerase chain reaction (PCR) and sequencing as conventional culture methods are lacking sensitivity regarding diagnosis of spontaneous bacterial peritonitis (SBP).

All patients with routinely performed ascitic fluid puncture and underlying liver cirrhosis are included in this study. Next generation sequencing (NGS) in ascitic fluid, skin swaps from puncture side and stool samples as well as conventional culture methods are performed to investigate the difference in the microbiome between patients with and without SBP.

ELIGIBILITY:
Inclusion Criteria:

* Underlying decompensated liver cirrhosis
* routinely performed ascitic fluid puncture
* informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with underlying liver cirrhosis and ascitic fluid that is routinley punctured.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Next generation sequencing results from ascitic fluid samples | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria